CLINICAL TRIAL: NCT00053456
Title: Stem Cell Mobilization For Improvement in Vascular Function and Myocardial Perfusion in Patients Undergoing Cardiac Rehabilitation
Brief Title: The Effect of Exercise on Stem Cell Mobilization and Heart Function in Patients Undergoing Cardiac Rehabilitation
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030086; 03-H-0086
Record Dates: First submitted 2003-01-30; First posted 2003-01-30 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Coronary Arteriosclerosis
Keywords: Endothelium; Nitric Oxide; Myocardial Ischemia; Exercise; Endothelial Progenitor Cells
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Motor Activity

SUMMARY:
This study will look at the effect of a cardiac rehabilitation exercise program on release of stem cells from the bone marrow and on heart function. Stem cells are primitive cells produced and released by the bone marrow, circulate in the bloodstream and develop into white blood cells, red blood cells and platelets. Some stem cells may also develop into other kinds of cells, including those that make up heart muscle, especially if the heart has been damaged or is not getting sufficient blood. Stem cells called endothelial progenitor cells (EPCs) are thought to form new blood vessels that can carry blood to areas of the heart muscle that are oxygen-deprived because of clogged arteries. Previous experiments have shown that some EPCs can be forced out of the bone marrow by exercise. This study will examine whether repeated exercise and lifestyle changes increase the number of EPCs released into the bloodstream and if these cells improve heart and blood vessel function.

Patients 21 years of age and older with coronary artery disease may be eligible for this study. Candidates will be screened with a medical history and physical examination, including a cardiovascular evaluation, and blood tests. The participants will be enrolled in a 2- to 3-month cardiac rehabilitation program that includes 24 to 36 60-minute sessions of exercise, plus instruction on lifestyle changes related to diet, stress management, and relaxation techniques. In addition, participants will undergo the following tests and procedures:

* Brachial reactivity study: This test measures how well the arteries widen. The patients rest for 30 minutes, and then an ultrasound device is placed over the artery just above the elbow. The device measures the size of the artery and blood flow through it before and after the patient is given a spray of nitroglycerin under the tongue.
* Blood tests for EPC levels and genetic testing: These measure EPCs and determine whether certain genes that may regulate EPC function are turned on or off. Genes are made up of DNA, the molecules that lead to the production of proteins by cells. Some of these proteins may be important in releasing EPCs from the bone marrow to travel in the bloodstream to the heart and repair blood vessels and muscle cells.
* Treadmill exercise testing: Patients exercise on a treadmill with continuous monitoring of the heartbeat and frequent measurements of oxygen saturation, using a finger clip device. The patient continues to exercise until moderate chest pain, shortness of breath, or fatigue develops.
* Questionnaire: Patients fill out a 15-minute questionnaire about their general physical and mental health status at the first and last visits to the clinic.
* Magnetic resonance imaging (MRI) of the heart: Patients who are eligible to undergo MRI have this test twice during the study, once before beginning the rehabilitation program and again after completing the program. The MRI shows heart function and blood flow in the heart. For this test, the patient lies on a stretcher inside a long narrow cylinder (the scanner). During the scan, the drug dipyridamole, which increases blood flow to the heart, is infused into a vein of the hand or arm. Another drug, gadolinium, is also infused to brighten the images produced.

DETAILED DESCRIPTION:
Exercise training has long been recommended as a means of improving cardiac function and reducing morbidity and mortality in patients with coronary artery disease (CAD). One mechanism of benefit may be through improved endothelial function and enhanced nitric oxide bioactivity. Such an effect may augment blood flow to exercising skeletal muscle and to the myocardium. In this regard, studies in both animals and humans have shown that frequent exercise improves endothelial function as well as blood flow to ischemic myocardium. Exercise-induced improvement in endothelial function is believed to result from up-regulation of endothelial nitric oxide synthase (eNOS) transcription due to repetitive shear stress associated with exercise. However, not all patients show improved endothelial function or myocardial perfusion despite compliant participation in cardiac rehabilitation programs. We hypothesize that endothelial function before and following structured exercise programs may be determined by the presence and function of endothelial progenitor cells (EPCs) that are released from the bone marrow and circulate in the blood stream. Thus, patients who have low baseline or post-exercise EPC levels or function may have limited capacity to improve endothelial function, exercise duration, and myocardial perfusion and function following participation in cardiac rehabilitation programs with repetitive exercise. On the other hand, patients with higher levels of EPCs at baseline or following repetitive exercise, with preserved capacity of EPCs to form endothelial cells, may show improved endothelial function, exercise duration, and myocardial perfusion and function as a result of repetitive exercise. The primary endpoint of this study will be improvement in endothelial function as determined by flow-mediated dilator responsiveness of the brachial artery at 2-3 months of repetitive exercise in the program compared with baseline measurements. Secondary endpoints include treadmill exercise duration and magnetic resonance imaging (MRI)-determined regional cardiac perfusion by gadolinium distribution during pharmacologic stress at 2-3 months compared with baseline measurements. EPCs will be identified by characteristic cell surface markers and by colony-forming ability at specific time-points of the study, with correlations determined between EPCs at baseline or the increase in EPCs following repetitive exercise, and the primary and secondary endpoints. We propose that patients most likely, and least likely, to benefit from a cardiac rehabilitation program may be identified on the basis of circulating EPCs.

ELIGIBILITY:
INCLUSION CRITERIA:

Adults older than 21 years.

Coronary artery disease established by angiography.

No myocardial infarction within 1 month.

Left ventricular ejection fraction greater than 30%.

No congestive heart failure symptoms within 2 months.

No medical condition that might prohibit safe participation in cardiac rehabilitation.

Subject understands protocol and provides written, informed consent in addition to willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

Significant structural heart disease (e.g. hypertrophic or dilated cardiomyopathy, valvular heart disease) as determined by echocardiography.

Angina pectoris that is prolonged in duration (greater than 20 minutes), or does not respond to nitroglycerin (2 tablets).

Subject physically unable to perform cardiac rehabilitation protocol due to neurologic or orthopedic conditions.

Hypersensitivity to organic nitrates.

Women of childbearing age unless recent pregnancy test is negative.

Lactating women.

Known hypersensitivity to dipyridamole or to gadolinium if patient eligible for MRI study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ades PA. Cardiac rehabilitation and secondary prevention of coronary heart disease. N Engl J Med. 2001 Sep 20;345(12):892-902. doi: 10.1056/NEJMra001529. No abstract available. PMID 11565523
- [Background] Belardinelli R, Georgiou D, Ginzton L, Cianci G, Purcaro A. Effects of moderate exercise training on thallium uptake and contractile response to low-dose dobutamine of dysfunctional myocardium in patients with ischemic cardiomyopathy. Circulation. 1998 Feb 17;97(6):553-61. doi: 10.1161/01.cir.97.6.553. PMID 9494025
- [Background] Bogle RG, Baydoun AR, Pearson JD, Mann GE. Regulation of L-arginine transport and nitric oxide release in superfused porcine aortic endothelial cells. J Physiol. 1996 Jan 1;490 ( Pt 1)(Pt 1):229-41. doi: 10.1113/jphysiol.1996.sp021138. PMID 8745290